CLINICAL TRIAL: NCT05365919
Title: The Family Talk Intervention in Clinical Practice When a Parent With Dependent Children is Severely Ill: An Effectiveness-implementation Study
Brief Title: Family Talk Intervention in the Context of Specialised Palliative Home Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ersta Sköndal University College (Other)
Collaborators: Forte (Industry)
Responsible Party: Principal Investigator, Malin Lövgren, Associate professor, Ersta Sköndal University College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Marie Cederschiöld University
Record Dates: First submitted 2022-03-04; First posted 2022-05-09 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Terminal Illness
Keywords: Specialised palliative care; Communication; Family Intervention
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: A cluster-randomized trial will be conducted at 12 homecare services (6 services=intervention, 6 services=control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will be offered to participate in the Family Talk Intervention
  Interventions: Other: Family Talk Intervention
- Standard support (No Intervention): The control group will receive standard support

INTERVENTIONS:
Other: Family Talk Intervention — FTI entails six meetings, with intervals of 1-2 weeks between meetings. Meetings 1-2 include only the parent(s) and focus on their experiences of the situation, as well as the consequences of the diagnosis for each family member. The parent(s) will formulate the goal of the intervention. Meeting 3: Interviews will be held with each child and includes the child's life situation. Meeting 4 includes the parent(s) and focuses on planning the family meeting. The children's thoughts and questions serve as a guide for the upcoming family meeting. Meeting 5 is a family meeting and consists of questions and issues raised earlier by the family members. Meeting 6 is a follow-up with all family members. The meeting is guided by the family members' needs, e.g., regarding communication and parenting. If the intervention is interrupted unexpectedly and cannot be finished as scheduled due to extraordinary circumstances, extra meetings are available (Meetings 7-11).
  Other Names: Beardslee's intervention
  Arms: Intervention

SUMMARY:
This intervention study aims to evaluate a psychosocial family based intervention in clinical practice, the Family Talk Intervention (FTI), for families with dependent children affected by life-threatening/life-limiting illness, when a parent is ill.

The study has an effectiveness implementation hybrid design where both the effects of FTI and the implementation process in clinical practice are examined.

DETAILED DESCRIPTION:
When a family with dependent children is affected by severe illness this affects the entire family. Still, there is little research evaluating support to such families. This intervention study aims to evaluate a psychosocial family based intervention in clinical practice, the Family Talk Intervention (FTI), for families with dependent children affected by life-threatening/life-limiting illness, when a parent is ill.

The study has an effectiveness implementation hybrid design where both the effects of FTI and the implementation process in clinical practice are examined. FTI will be carried out as a cluster randomized trial at 12 clinics in specialized palliative homecare (6 units=intervention, 6 units=control).

All social workers at these clinics will receive education and training in FTI in 2021. From 2022, FTI will be offered to families cared for at these care contexts.

FTI is manual-based and consists of 6 meetings with the families (together and individually) and is led by the FTI-educated social workers. The aim of FTI are to support the family in talking about illness-related subjects (e.g. prognosis, stress), support parenting, and support the family in identifying their strengths and how to best use them.

FTI will be evaluated through surveys and interviews with families before FTI/baseline and after completed intervention (3 and 6 months after baseline). Further, social workers will be invited to compete questionnaires and take part in focus groups about their experiences of FTI.

The research group has conducted pilot-studies on FTI in these contexts with positive results. The present study allows us to take a further step in the evaluation of FTI- evaluate FTI under real conditions.

ELIGIBILITY:
Inclusion Criteria:

* Families affected by a life-threatening or life-limiting illness and have dependent children, ill or health aged 0-19 years and
* Enrolled in specialized palliative home care
* At least two family members have accepted to participate

Exclusion Criteria:

-

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in family Communication over time. Family Adaptability and Cohesion Scale IV | Six months
  Measures in self-rated family communication which is the primary outcome of the intervention

SECONDARY OUTCOMES:
Changes in self-rated resilience. Resilience Scale (RS-14) ((Resilience Scale for Children (RS-10)). | Six months
  Measures self-rated resilience in adults and children
Changes in self-rated grief. Prolonged Grief Disorder (PG-12/PG-13). | Six months
  An instrument to screen for pathologic forms of grief before and after an expected death
Changes in self-rated anxiety. Generalized Anxiety Disorder (GAD) | Six months
  Measures symptoms of anxiety
Changes in The Strengths and Difficulties Questionnaire (SDQ) | Six months
  Measures self-rated strengths and difficulties. Has a proxy version for children
Changes in self-perceived parenting skill. Parental Skills Checklist (PSC) | Six months
  Measures self-rated parenting abilities
Changes in factors needed for successful implementation.The Swedish Normalization Process Theory Measure (S-NoMAD) | Six months
  For the implementation research. Characterizes and explains key mechanisms that promote and inhibit the implementation, embedding and integration of new health techniques, technologies and other complex interventions.
Changes in perception of organizational context. Alberta Context Tool (ACT) | Six months
  For the implementation research. Measures organizational context for use in complex healthcare settings.

CONTACTS AND LOCATIONS:
Overall Officials: Malin Lövgren, PhD, Principal Investigator — Marie Cederschiölds University College
Locations (1):
- Marie Cederschiöld Unicersity College, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thermaenius I, Holm M, Arestedt K, Udo C, Alvariza A, Lundberg T, Wallin L, Lovgren M. Implementing the Family Talk Intervention among families with a severely ill parent or child with palliative care needs- a longitudinal study of the perspectives of hospital social workers. Front Health Serv. 2025 Jun 13;5:1527431. doi: 10.3389/frhs.2025.1527431. eCollection 2025. PMID 40584244